CLINICAL TRIAL: NCT05077163
Title: Renal Assessment of Patients With Acute Renal Failure During Severe COVID-19
Brief Title: Patients With Acute Renal Failure During Severe COVID-19
Acronym: IR-EST-POSTCOV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8039
Record Dates: First submitted 2021-10-13; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Renal Failure Chronic
Keywords: COVID-19; SARS-COV-2; Renal failure
MeSH Terms: conditions — Renal Insufficiency, Chronic; COVID-19; Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The occurrence of renal failure during severe forms of COVID-19 is common (20-35% of patients treated in intensive care) and associated with an unfavorable short-term prognosis, but the medium-term renal outcome is not is not known.

The aim of the study is to establish the frequency of chronic kidney failure after AKI KDIGO 2 and 3 occurring during severe COVID-19 in intensive care.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Subject hospitalized in an intensive care unit, Strasbourg, Nancy or Reims hospitals, for severe COVID-19 between February 1, 2020 and July 31, 2020.
* Having presented acute renal failure KDIGO 2 (assessed on a doubling of serum creatinine compared to the patient's reference values) or 3 (serum creatinine greater than 3 times the patient's reference, or anuria, or any recourse to extra-purification renal)
* Having left hospital alive after initial treatment for COVID-19
* Subject not having expressed his opposition, after information, to the reuse of his data for the purposes of this research.

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Subject under guardianship or guardianship
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - Major subject hospitalized in an intensive care unit, Strasbourg, Nancy or Reims Hospitals, for severe COVID-19 between February 1, 2020 and July 31, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of renal development in patients with acute renal failure during severe COVID-19 | Files analysed retrospectively from February 01, 2020 to July 31, 2020 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Bruno MOULIN, MD, PhD, Principal Investigator — Service de Néphrologie et Transplantation - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Néphrologie et Transplantation - Hôpitaux Universitaires de Strasbourg, Strasbourg, France